CLINICAL TRIAL: NCT01532349
Title: Cholecalciferol as a Modifier of Serum Hepcidin in Children With Chronic Kidney Disease
Brief Title: Vitamin D as a Modifier of Serum Hepcidin in Children With Chronic Kidney Disease
Acronym: D-fense
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00066175; 1K23DK084116-01A2 (NIH)
Record Dates: First submitted 2012-02-08; First posted 2012-02-14 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: chronic kidney disease; anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 400 IU vitamin D (Active Comparator): Children will be randomly allocated to receive cholecalciferol supplementation 400 IU/day (2,800 IU/weekly), which is the recommended dietary allowance. Study participants will be prescribed any clinically indicated additional cholecalciferol supplementation once the 3-month laboratory measures have been obtained, based on serum 25D levels at the end of the study period.
  Interventions: Drug: Cholecalciferol
- 4000 IU vitamin D (Active Comparator): Children will be randomly allocated to receive cholecalciferol supplementation 4000 IU/day (28,000 IU weekly) according to the KDOQI recommended supplementation for children with mild 25D deficiency. Study participants will be prescribed any clinically indicated additional cholecalciferol supplementation once the 3-month laboratory measures have been obtained, based on serum 25D levels at the end of the study period.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Children will be randomly allocated to receive either cholecalciferol supplementation 4000 IU per day 400 IU/day. We are proposing a supplementation dose of 4000 IU/day in children with CKD, which is considered a safe dose by KDOQI standards; vitamin D2 doses as high as 10,000 IU/day have been given to French patients with CKD for > 1 year with no evidence of vitamin D toxicity. Cholecalciferol will be provided in both tablet and liquid form, based on the ability to tolerate and preference of the subject. Participants will be monitored for signs of 25D toxicity (hypercalcemia, hyperphosphatemia, hypercalciuria) during the follow up period of 1 month and 3 months from baseline.
  Other Names: tablet: National Vitamin Company, Casa Grande, AZ; liquid: Enfamil® D-Vi-Sol™ Drops

SUMMARY:
This research is being done to study the effectiveness of vitamin D (cholecalciferol) to modify hepcidin levels in children with chronic kidney disease (CKD). Anemia is a common problem in children with CKD. Anemia is when the body does not have enough healthy red blood cells. Hepcidin is a protein in the blood which interferes with the body's production of red blood cells. This study will see if vitamin D lowers hepcidin levels in children and young adults with CKD. If so, it could be used as an additional treatment for anemia in these children, in addition to the current therapies already in use including iron supplements and erythropoietin. People between the ages of 1 and 21 with CKD may be considered for this study.

DETAILED DESCRIPTION:
Vitamin D Supplementation is a practical and inexpensive intervention which is safe, readily available and clinically indicated. Substantial recent evidence suggests vitamin D may modify inflammatory pathways in CKD. There is a high probability of benefit and a low probability of harm for this easily modifiable factor. 25D levels can be effectively modified through oral supplementation with cholecalciferol. To the best of our knowledge, no studies examining the effects of oral cholecalciferol supplementation on hepcidin levels have been conducted in children with either CKD or other diseases.

We will conduct a randomized open-label controlled trial of oral cholecalciferol supplementation in children aged 1-21 years with stage 2-5 (pre-dialysis) CKD receiving regular nephrology follow-up at a tertiary-care children's hospital (Johns Hopkins Children's Center). The intervention model will be parallel assignment. Children will be randomly allocated to receive either cholecalciferol supplementation 4000 IU per day (28,000 IU weekly) according to the KDOQI recommended supplementation for children with mild 25D deficiency, or will be treated with 400 IU/day (2,800 IU/weekly), which is the recommended dietary allowance.(1) Allocation will be double-blinded to prevent knowledge of allocation status affecting interpretation of results. Study participants will be prescribed any clinically indicated additional cholecalciferol supplementation once the 3-month laboratory measures have been obtained, based on serum 25D levels at the end of the study period.(1) We are proposing a supplementation dose of 4000 IU/day in children with CKD, which is considered a safe dose by KDOQI standards; vitamin D2 doses as high as 10,000 IU/day have been given to French patients with CKD for > 1 year with no evidence of vitamin D toxicity.(2) 25D levels between 40 and 80 are indicative of "sufficiency", and a safe upper limit of intake, in which the risk of hypercalcemia is negligible, has been defined as 10,000 IU/day.(3, 4) Cholecalciferol will be provided in both tablet (vitamin D 2000 IU tablets and 400 IU tablets, National Vitamin Company, Casa Grande, AZ) and liquid (Enfamil® D-Vi-Sol™ Drops, 400 IU per mL) form, based on the ability to tolerate and preference of the subject.

Participants will be monitored for signs of 25D toxicity (hypercalcemia, hyperphosphatemia, hypercalciuria) during the follow up period of 1 month and 3 months from baseline.

Data Safety Monitoring Board will review serum calcium, phosphorus, and urine calcium:creatinine ratio values at the one month visit; if subjects show evidence of hypercalcemia or hyperphosphatemia (serum values > upper limit of normal, age-specific values, see Table 3 below), study drug will be discontinued.(3) If subjects demonstrate evidence of hypercalciuria (urine calcium:cr ratio > 0.6 in 1-2 year olds or > 0.2 in > 2 year olds) study drug will be discontinued.(5) In addition, if 25-hydroxy vitamin D levels > 80 ng/mL are reached, the study drug will be discontinued. In any subject in whom study drug is discontinued, the 3-month laboratory data will still be collected.

In the case of hypoalbuminemia (serum albumin < 3.5 g/dL) corrected total serum calcium will be calculated using the formula: Corrected calcium (mg/dL) = serum calcium (mg/dL) + 0.8 (4 - serum albumin [g/dL])(2) Standardized blood pressure measurement will include three manual BP measurements conducted after five minutes of rest with an aneroid sphygmomanometer, at least 30 seconds apart.

1. KDOQI Work Group. KDOQI clinical practice guideline for nutrition in children with CKD: 2008 update. executive summary. Am J Kidney Dis. 2009 Mar;53(3 Suppl 2):S11-104.
2. KDOQI clinical practice guidelines for bone metabolism and disease in children with chronic kidney disease. Am J Kidney Dis. 2005;46(Supplement 1):S1-S122.
3. Querfeld U, Mak RH. Vitamin D deficiency and toxicity in chronic kidney disease: In search of the therapeutic window. Pediatr Nephrol. 2010 Jun 22.
4. Shroff R, Knott C, Rees L. The virtues of vitamin D--but how much is too much? Pediatr Nephrol. 2010 Sep;25(9):1607-20.
5. Kruse K, Kracht U, Kruse U. Reference values for urinary calcium excretion and screening for hypercalciuria in children and adolescents. Eur J Pediatr. 1984 Nov;143(1):25-31.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stage 2-5 Chronic Kidney Disease (estimated glomerular filtration rate [GFR] between 15 and < 90 ml/min/1.73m2) based on the new bedside Schwartz formula estimation using serum creatinine and height [height in cm x 0.413/serum creatinine]
* 1-21 years of age
* Willingness and ability to provide informed consent and assent

Exclusion Criteria:

* Children less than 1 year of age (in whom risk of vitamin D toxicity may be increased) or greater than 21 years at time of study screening
* Children with a documented history of hypercalcemia or nephrolithiasis
* Children with GI tract discontinuity (ostomy)
* Current pregnancy or pregnancy within the last 12 months
* Children with known anemia-related disorders including sickle cell anemia, thalassemia
* Children with severe 25D deficiency (< 5 ng/mL) likely to be associated with severe morbidity and requiring prompt high dose vitamin D supplementation, or with 25D levels > 60 ng/mL which could be associated with increased risk of vitamin D toxicity

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Atkinson, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 400 IU Vitamin D | 4000 IU Vitamin D
Started | 17 | 17
Completed | 15 | 12
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- 400 IU Vitamin D: Children were randomly allocated to receive cholecalciferol supplementation 400 IU/day (2,800 IU/weekly), which is the recommended dietary allowance. Study participants will be prescribed any clinically indicated additional cholecalciferol supplementation once the 3-month laboratory measures have been obtained, based on serum 25D levels at the end of the study period.
- 4000 IU Vitamin D: Children were be randomly allocated to receive cholecalciferol supplementation 4000 IU/day (28,000 IU weekly) according to the KDOQI recommended supplementation for children with mild 25D deficiency. Study participants will be prescribed any clinically indicated additional cholecalciferol supplementation once the 3-month laboratory measures have been obtained, based on serum 25D levels at the end of the study period.
- Total: Total of all reporting groups
Arm/Group | 400 IU Vitamin D | 4000 IU Vitamin D | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 15 | 28
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (6.3) | 10.8 (5.5) | 10.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Hepcidin With Vitamin D Intervention for Children With Chronic Kidney Disease
Description: The null hypothesis to be tested is that Vitamin D supplementation will not be associated with a decrease in serum hepcidin over the study period. Statistical analysis will be performed as intention-to-treat.
Time Frame: change from baseline to up to three months
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- 400 IU Vitamin D: Children were randomly allocated to receive cholecalciferol supplementation 400 IU/day (2,800 IU/weekly), which is the recommended dietary allowance. Study participants will be prescribed any clinically indicated additional cholecalciferol supplementation once the 3-month laboratory measures have been obtained, based on serum 25D levels at the end of the study period.
  Serum hepcidin was the primary outcome variable and was quantified at all visits.
- 4000 IU Vitamin D: Children were be randomly allocated to receive cholecalciferol supplementation 4000 IU/day (28,000 IU weekly) according to the KDOQI recommended supplementation for children with mild 25D deficiency. Study participants will be prescribed any clinically indicated additional cholecalciferol supplementation once the 3-month laboratory measures have been obtained, based on serum 25D levels at the end of the study period.
  Serum hepcidin was the primary outcome variable and was quantified at all visits.
Arm/Group | 400 IU Vitamin D | 4000 IU Vitamin D
Number analyzed (Participants) | 15 | 12
ng/ml | 48.2 [38 to 63] | 75.4 [38.6 to 123.12]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | 400 IU Vitamin D | 4000 IU Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 5/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 IU Vitamin D (N=17) | 4000 IU Vitamin D (N=17)
Hyperphosphatemia (Renal and urinary disorders) | 0 (0) | 1 (1) — (serum phosphorus > 6.5 mg/dl in 1-5 year-olds, > 5.8 in 6-12 year-olds, or > 4.5 in 13-20 year-olds
Hypervitaminosis D (Endocrine disorders) | 0 (0) | 3 (3) — 25hydroxyvitamin D levels > 60 ng/ml were noted at the 4-week visit
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) — Kidney stone incidentally noted on imaging

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No